CLINICAL TRIAL: NCT02947945
Title: Open-Label, to Evaluate the Efficacy and Safety of Reslizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis (EGPA) Study: RITE Study
Brief Title: Reslizumab in the Treatment of Eosinophilic Granulomatosis With Polyangiitis (EGPA) Study
Acronym: RITE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Michael Wechsler, Prinicipal Investigator, National Jewish Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-3025
Record Dates: First submitted 2016-10-17; First posted 2016-10-28 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — reslizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Other): all subjects will receive the study medication- reslizumab.
  Interventions: Drug: Reslizumab

INTERVENTIONS:
Drug: Reslizumab — All subjects will receive Reslizumab
  Other Names: Cinqair

SUMMARY:
Reslizumab is a type of medicine called a monoclonal antibody that is made in the research clinic; it works by blocking a specific protein in the body called interleukin-5. The study medicine, reslizumab, is not yet approved for doctors to treat patients with EGPA. It is considered an experimental drug in this study.

DETAILED DESCRIPTION:
This study is open-label which means that all subjects will receive the study medication. The study medicine - reslizumab - will be given to the participants in addition to the medicines they are already taking to treat their EGPA such as oral steroids (e.g. prednisone) and medicines that reduce the activity of their immune system (the study doctor will tell the participants which medications these are) - this is what is meant by 'standard of care' and can vary in different countries. Drugs that are sometimes used (i.e., 'standard of care') to reduce the activity of the immune system in EGPA (in addition to oral steroids) include azathioprine, methotrexate, mycophenolate mofetil and cyclophosphamide. Information about how the study drug affects the human body and health will be collected through a number of tests, procedures and questions.

The study medicine, reslizumab, will be given to the participants at a dose of 3mg/kg intravenously (within a vein) every four weeks for 28 weeks for a total of 7 treatments. During the treatment phase of this study, a study staff member will call the participants every two weeks to see how they are doing, what medications they are taking, and if they are able to decrease their steroid use. The study is a total of 11 study visits in a 44 week time period. Everyone who takes part in the study will continue to receive his/her existing treatments for EGPA (although the dose of oral steroids may be reduced during the study).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Gender and Age: Male or female subjects >18 years old
* EGPA diagnosis: subjects who have been diagnosed with EGPA for at least 6 months based on the history or presence of: asthma plus eosinophilia (>1.0x109/L and/or >10% of leucocytes) plus at least two of the following additional features of EGPA:

  * A biopsy showing histopathological evidence of eosinophilic vasculitis, or perivascular eosinophilic infiltration, or eosinophil-rich granulomatous inflammation;
  * Neuropathy, mono or poly (motor deficit or nerve conduction abnormality);
  * Pulmonary infiltrates, non-fixed;
  * Sino-nasal abnormality;
  * Cardiomyopathy (established by echocardiography or MRI);
  * Glomerulonephritis (haematuria, red cell casts, proteinuria);
  * Alveolar haemorrhage (by bronchoalveolar lavage);
  * Palpable purpura;
  * ANCA positive (MPO or PR3).
* Subjects who have received a cyclophosphamide (CYC) induction regimen may be included a minimum of 2 weeks after the last dose of daily oral CYC, or 3 weeks after the last dose of pulsed IV CYC prior to visit 1, if their total WBC is ≥4x109/L prior to visit 1.
* Subjects who have received a methotrexate, azathioprine, or mycophenolate mofetil induction regimen may be included if on a stable dose for at least 4 weeks prior to visit 1.
* Corticosteroid therapy: Subject must be on a stable dose of oral prednisolone or prednisone of ≥5 mg/day for at least 4 weeks prior to visit 1.
* Immunosuppressive therapy: If receiving immunosuppressive therapy (including methotrexate, azathioprine, or mycophenolate mofetil, but excluding restricted medications below) the dosage must be stable for the 4 weeks prior to visit 1 and during the study (dose reductions for safety reasons will be permitted).
* Female subjects: To be eligible for entry into the study, females of childbearing potential (FCBP) must commit to consistent and correct use of an acceptable method of birth control beginning with consent, for the duration of the trial.

Exclusion Criteria:

* Hypereosinophilic Syndrome
* Wegener's Granulomatosis
* Malignancy
* Parasitic disease
* Pregnant or nursing
* If female and of child-bearing potential, must have negative pregnancy test and must adhere to acceptable method of contraception (with <1% failure rate) during the study and for four months after the study.
* Any other medical illness that precludes study involvement
* Patients who are currently receiving or have previously received reslizumab or any other type of anti-interleukin therapy (i.e. mepolizumab, lebrikizumab etc.) within the last three months.
* Taking cyclophosphamide
* Any patients with a known hypersensitivity to reslizumab or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Document the safety of reslizumab therapy in patients with EGPA | up to 12 months
  All adverse events will be reported to the sponsor and the IRB in accordance with the policy of National Jewish Health and the FDA. Adverse events will be recorded on Case Report Forms as non-serious or serious events (DAEs). Serious adverse events, whether or not considered related to the investigational drug, will be recorded on the Serious Adverse Event form and faxed to the IRB and the sponsor as soon as site personnel are aware of the event. Every attempt will be made to collect discharge summaries for each hospitalization should they occur to provide further details.

SECONDARY OUTCOMES:
Demonstrate the steroid sparing effect of reslizumab therapy by titrating corticosteroid dosage | up to 12 months
  Goal is to demonstrate the steroid sparing effect of reslizumab therapy by titrating corticosteroid dosage while using this anti-IL-5 therapy or to reduce the rate of EGPA exacerbations during the study period. Change in steroid dose will be assessed by comparing the corticosteroid dose of subjects at the end of the steroid stable phase and compare to steroid dose at the end of the treatment period. Change in the rate of exacerbations will be assessed by comparing the rate of exacerbations during the study period with the rate during the washout and safety-monitoring period as well as with the self-reported rate of exacerbations from the year prior to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wechsler, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manka LA, Guntur VP, Denson JL, Dunn RM, Dollin YT, Strand MJ, Wechsler ME. Efficacy and safety of reslizumab in the treatment of eosinophilic granulomatosis with polyangiitis. Ann Allergy Asthma Immunol. 2021 Jun;126(6):696-701.e1. doi: 10.1016/j.anai.2021.01.035. Epub 2021 Feb 4. PMID 33548468